CLINICAL TRIAL: NCT04711902
Title: A Phase III Randomized, Double-blind, Placebo Controlled, Multicenter, Bridging Study of Subcutaneous Secukinumab, to Demonstrate Efficacy After Sixteen Weeks of Treatment and to Assess Safety, Tolerability and Long-term Efficacy Follow-up to One Year in Chinese Subjects With Active Psoriatic Arthritis
Brief Title: Study of Efficacy and Safety of Secukinumab in Chinese Subjects With Active PsA Compared to Placebo.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2367
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Psoriatic Arthritis
Keywords: PsA; immune-mediated chronic inflammatory disease; spondylarthritis; SpA; inflammatory musculoskeletal disease; China bridging study; AIN457; secukinumab
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylarthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Participants received 150 mg dose (dose level 1) of Secukinumab
  Interventions: Drug: AIN457
- Arm 2 (Placebo Comparator): Participants received Placebo of the study drug.
  Interventions: Other: Secukinumab Placebo
- Arm 3 (Active Comparator): Participants who received Placebo and switched to dose level 1 (150 mg) of secukinumab.
  Interventions: Drug: AIN457; Other: Secukinumab Placebo
- Arm 4 (Active Comparator): Participants who received Placebo and switched to dose level 2 (300 mg) of secukinumab.
  Interventions: Drug: AIN457; Other: Secukinumab Placebo

INTERVENTIONS:
Drug: AIN457 — Secukinumab 150 mg was supplied in 1.0 mL prefilled syringe, administered via subcutaneous injection
  Other Names: Secukinumab
  Arms: Arm 1; Arm 3; Arm 4
Other: Secukinumab Placebo — Secukinumab placebo was supplied in 1.0 mL prefilled syringe, administered via subcutaneous injection
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
The purpose of this study was to assess the efficacy and safety of secukinumab in Chinese participants with active Psoriatic arthritis (PsA ) compared to placebo.

DETAILED DESCRIPTION:
This study used a randomized, double-blind, placebo-controlled, parallel-group design.

A screening period running up to 10 weeks before randomization was used to assess participant eligibility followed by 52 weeks of treatment.

A follow-up visit was done 12 weeks after last study treatment administration for all participants, regardless of whether they completed the entire study as planned or discontinued prematurely.

At Baseline, the patients fulfilling the inclusion criteria were randomized to one of the following two groups.

Group 1 : Secukinumab Dose level 1 s.c. at BSL, Week 1, 2, 3, 4, 8, and 12 Group 2 : Secukinumab Placebo s.c. at BSL, Week 1, 2, 3, 4, 8, and 12.

At Week 16, participants in Group 1 and Group 2 were to be re-randomized separately in a 1:1 ratio to receive secukinumab 150 mg or secukinumab 300 mg.

The duration of the entire treatment period was 52 weeks.

The primary objective was to demonstrate the treatment effect of secukinumab in Chinese subjects with active PsA by assessing American College of Rheumatology rresponse 20 (ACR20 response) rates at Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed.
* Chinese male or non-pregnant, non-lactating Chinese female participants at least 18 years of age.
* Diagnosis of PsA classified by Classification of Psoriatic Arthritis (CASPAR) criteria and with symptoms for at least 6 months with moderate to severe Psoriatic arthritis (PsA).
* Rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) antibodies negative at screening.
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis or a documented history of plaque psoriasis.
* Participants on Methotrexate (MTX) must be on folic acid supplementation at randomization.
* Participants who are on a DMARD other than MTX must discontinue the DMARD 4 weeks prior to randomization visit except for leflunomide, which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine washout has been performed.

Exclusion Criteria:

* Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician
* Participants taking high potency opioid analgesics (e.g., methadone, hydromorphone, morphine).
* Previous exposure to secukinumab or other biologic drug directly targeting interleukin- 17 (IL-17) or IL-17 receptor
* Participants who have ever received biologic immunomodulating agents except for those targeting Tumor necrosis factor alpha (TNFα).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective contraception during the entire study (during the entire study).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- China (12):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhuzhou, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the 1st 16 weeks of study, the 41 participants enrolled were randomized to 2 groups: 1 group received secukinumab 150 mg & the other received placebo. At week 16, the participants were re-randomized within each group for a total of 4 groups. Within the secukinumab group, 1 group continued to receive secukinumab 150 mg while the other half received secukinumab 300 mg. In the Placebo group, 1 group switched to secukinumab 150 mg while the other half switched to secukinumab 300 mg.
Pre-assignment Details: This study was conducted in 12 centers in China.
Groups:
- Secukinumab 150 mg (Group 1): Participants received 150 mg dose (dose level 1) of Secukinumab
- Placebo of Study Drug (Group 2): Participants received Placebo of the study drug
- Secukinumab 150 mg to Secukinumab 150 mg (2nd Randomization): Participants who had previously received Secukinumab 150 mg dose (dose level 1) continued receiving 150 mg dose (dose level 1) of Secukinumab
- Secukinumab 150 mg to Secukinumab 300 mg (2nd Randomization): Participants who had previously received Secukinumab 150 mg dose (dose level 1) now received 300 mg dose (dose level 2) of Secukinumab
- Placebo to Secukinumab 150 mg (2nd Randomization): Participants who had previously received Placebo switched to Secukinumab 150 mg (dose level 1)
- Placebo to Secukinumab 300 mg (2nd Randomization): Participants who had previously received Placebo switched to Secukinumab 300 mg (dose level 2)
Period: Treatment Period 1 (1st 16 Weeks)
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2) | Secukinumab 150 mg to Secukinumab 150 mg (2nd Randomization) | Secukinumab 150 mg to Secukinumab 300 mg (2nd Randomization) | Placebo to Secukinumab 150 mg (2nd Randomization) | Placebo to Secukinumab 300 mg (2nd Randomization)
Started | 20 | 21 | 0 | 0 | 0 | 0
Completed | 20 | 21 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (From Week 16)
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2) | Secukinumab 150 mg to Secukinumab 150 mg (2nd Randomization) | Secukinumab 150 mg to Secukinumab 300 mg (2nd Randomization) | Placebo to Secukinumab 150 mg (2nd Randomization) | Placebo to Secukinumab 300 mg (2nd Randomization)
Started | 0 | 0 | 10 | 10 | 10 | 11
Discont. From Treatment Before Week 52 | 0 | 0 | 0 | 0 | 1 | 0
Completed Study Treatment | 0 | 0 | 10 | 10 | 9 | 11
Completed | 0 | 0 | 8 | 10 | 10 | 11
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Participant decision | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set: All participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2) | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (9.70) | 45.7 (10.46) | 44.0 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 7 | 16 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: ACR20 Response at Week 16
Description: Assessed the efficacy of secukinumab relative to placebo at week 16 using Non-responder imputation (NRI) and based on the percentage of participants achieving an ACR20 response (ACR = American College of Rheumatology). ACR20 response criteria is response ≥ 20% improvement based on:
  Swollen Joint Count (SJC)/Tender Joint Count (TJC), Patient's global assessment of disease activity (PaGA) (Visual Analog Scale (VAS)), Physician's global assessment of disease activity (PhGA) (VAS), Patient's assessment of PsA pain intensity (VAS), Health Assessment Questionnaire - Disability Index (HAQ-DI), and High-sensitivity C-reactive protein (hsCRP) or Erythrocyte sedimentation rate (ESR).
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): All participants from the randomized set to whom study treatment had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 20 | 21
Participants | 14 | 6
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Regression, Logistic; Marginal difference = 39.91, 95% CI 2-sided [10.87 to 68.95]

2. Secondary Outcome: ACR50 Response at Week 16
Description: To assess the effect of secukinumab versus placebo on the composite endpoint ACR50 response and based on the percentage of participants achieving an ACR50 response at Week 16 using NRI. ACR50 response criteria is response ≥ 50% improvement based on: Swollen Joint Count (SJC)/Tender Joint Count (TJC), Patient's global assessment of disease activity (PaGA) (VAS), Physician's global assessment of disease activity (PhGA) (VAS), Patient's assessment of PsA pain intensity (VAS), HAQ-DI, and hsCRP or ESR.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): All participants from the randomized set to whom study treatment had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 20 | 21
Participants | 3 | 1
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Regression, Logistic; Marginal difference = 11.86, 95% CI 2-sided [-7.18 to 30.91]

3. Secondary Outcome: Change From Baseline in DAS28-CRP Scores Using Mixed Model Repeated Scores (MMRM) at Week 16
Description: To assess the effect of secukinumab versus placebo on change from BSL in DAS28-CRP. The assessment is based on the reduction in DAS28-CRP score.
  The DAS28 is a measure of disease activity based on Swollen and Tender Joint Counts, ESR or CRP and the Patient Global Assessment of Disease Activity. The range of DAS28 score is 0-10. Higher score means more active disease. Negative change from baseline indicates a favorable outcome.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): All participants from the randomized set to whom study treatment had been assigned. This is subset of participants from the randomized set to whom study treatment had been assigned and had a valid value of the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 18 | 20
scores on a scale | -1.47 (0.206) | -0.37 (0.200)
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Mixed Models Analysis; Mixed model repeated measures (MMRM) = -1.10, 95% CI 2-sided [-1.68 to -0.52]

4. Secondary Outcome: Change From Baseline in PASDAS Scores Using MMRM at Week 16
Description: To assess the the effect of secukinumab versus placebo on change from Baseline in PASDAS. Assessment was based on reduction in PASDAS score.
  PASDAS is a measure of disease activity based on Patient reported measures (excluding mental component score (MCS) of the medical outcomes survey Short Form-36 (SF-36-PCS)), skin, peripheral joint counts (Tender and Swollen joint counts), Dactylitis (LDI), Enthesitis (LEI), acute phase response (CRP) and Patient & Physician global VAS scores. The range of PASDAS is 0-10. Higher score means more active disease. Negative change from baseline indicates a favorable outcome.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 18 | 20
scores on a scale | -2.20 (0.245) | -0.55 (0.237)
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Mixed Models Analysis; Mixed model repeated measures (MMRM) = -1.65, 95% CI 2-sided [-2.35 to -0.94]

5. Secondary Outcome: Change From Baseline in SF36-PCS Scores Using MMRM at Week 16
Description: To assess the effect of secukinumab versus placebo on change from Baseline in SF-36 PCS.
  The SF-36 is a widely used and extensively studied instrument to measure HRQoL among healthy participants and participants with acute and chronic conditions. Two overall summary scores, the Physical Component Score (PCS) and the Mental Component Score (MCS) also can be computed. SF36-PCS was used in this study. The range of SF36-PCS score is 0-100. Higher score means better health status. Negative change from baseline indicates a unfavorable outcome.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 19 | 21
scores on a scale | 4.28 (1.154) | 0.08 (1.113)
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Mixed Models Analysis; Mixed model repeated scores (MMRM) = 4.20, 95% CI 2-sided [0.94 to 7.46]

6. Secondary Outcome: Change From Baseline in HAQ-DI Scores Using MMRM at Week 16
Description: To assess the effect of secukinumab versus placebo on change from Baseline in HAQ-DI. Assessment was based on improvement in HAQ-DI PCS scores.
  The HAQ-DI© is one of the most widely used measures to assess the long-term influence of chronic disease on a participant's level of functional ability and activity restriction, and calculated based on HAQ-DI questionnaire. There are 20 questions in eight categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The range of score is 0-3. Higher score means more severe disability. Negative change from baseline indicates a favorable outcome.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg (Group 1) | Placebo of Study Drug (Group 2)
Number analyzed (Participants) | 19 | 21
scores on a scale | -0.31 (0.065) | 0.09 (0.063)
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group 1) vs Placebo of Study Drug (Group 2); Test type: Other — estimation and confidence interval; Mixed Models Analysis; Mixed model repeated measures (MMRM) = -0.40, 95% CI 2-sided [-0.58 to -0.21]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study medication (on-treatment), up to approx. 52 weeks.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Any AIN457 150 mg: Participants who received Secukinumab 150 mg dose (dose level 1) at any point during the trial.
- Any AIN457 300 mg: Participants who received Secukinumab 300 mg dose (dose level 2) at any point during the trial.
- Any AIN457: Participants who received Secukinumab, regardless of dose, at any point during the trial.
- Placebo: Participants who received Placebo at any point during the trial.
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/21 | 0/41 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/21 | 1/41 | 0/21
Other Adverse Events (participants affected / at risk) | 27/30 | 16/21 | 37/41 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=30) | Any AIN457 300 mg (N=21) | Any AIN457 (N=41) | Placebo (N=21)
Cataract (Eye disorders) | 0 | 1 | 1 | 0
Epiretinal membrane (Eye disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=30) | Any AIN457 300 mg (N=21) | Any AIN457 (N=41) | Placebo (N=21)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 1 | 0
Retinoschisis (Eye disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Discomfort (General disorders) | 1 | 0 | 1 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2 | 5 | 0
COVID-19 (Infections and infestations) | 4 | 5 | 9 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 3 | 2 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 1 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram high voltage (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 1
Glucose urine present (Investigations) | 0 | 1 | 1 | 1
Protein urine present (Investigations) | 1 | 0 | 1 | 0
Total bile acids increased (Investigations) | 1 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 0
Urinary occult blood positive (Investigations) | 1 | 0 | 1 | 0
Weight increased (Investigations) | 3 | 0 | 3 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 0 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 3 | 9 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 4 | 9 | 2
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT04711902/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT04711902/SAP_001.pdf